CLINICAL TRIAL: NCT01941953
Title: Phase II Study of Metformin and 5-fluorouracil in Patients With Advanced Colorectal Cancer Previously Treated With Oxaliplatin and Irinotecan Based Chemotherapy.
Brief Title: Metformin and 5-fluorouracil for Refractory Colorectal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Vanessa C Miranda, Fellow in Clinical Oncology, Instituto do Cancer do Estado de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 273/12
Record Dates: First submitted 2013-09-04; First posted 2013-09-13 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metformin; Metastatic Colorectal Cancer; Fluorouracil
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metformin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin and Flourouracil (Experimental)
  Interventions: Drug: Metformin and Fluorouracil

INTERVENTIONS:
Drug: Metformin and Fluorouracil — metformin 850mg PO BID plus 5FU 425mg/m2 + leucovorin 50mg IV weekly

SUMMARY:
This is a phase II trial to evaluate efficacy and safety of Metformin and Fluorouracil in patients with metastatic colorectal cancer (CRC) who have progressed after Oxaliplatin and Irinotecan based chemotherapy.

DETAILED DESCRIPTION:
Primary Outcomes Measures:

- Disease control Rate at 8 weeks according to RECIST 1.1 (Tumor response was defined as the percentage of patients with complete response, partial response or stable disease as best overall response).

Secondary Outcome Measures:

* Progression-free Survival
* Overall Survival
* Adverse Events (assessed according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0)

ELIGIBILITY:
Inclusion Criteria

* Histological diagnosis of metastatic colorectal adenocarcioma previously treated with at least two lines of chemotherapy (oxaliplatin and irinotecan regimens) if mutated KRAS or treated with at least 3 lines of chemotherapy (oxaliplatin, irinotecan and cetuximab) if KRAS wild type.
* Disease progression according to radiological or clinical assessment.
* Measurable disease.
* ECOG Performance 0-1.
* Age above 16 years.
* Normal organic function as defined for the following criteria:

  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 times the upper normal limit of the local laboratory (LSN-LL);
  * Total serum bilirubin ≤ 2.0 x ULN-LL;
  * Absolute neutrophil count ≥ 1,500 / mm3;
  * Platelet count ≥ 100,000 / mm3;
  * Hemoglobin ≥ 8.0 g / dl;
  * Serum creatinine ≤ 1.5 x ULN-LL
* Written informed consent before enrollment

Exclusion Criteria

* Diabetic patients taking metformin.
* Patients already treated with mTOR inhibitors.
* Hypersensitivity to metformin, renal or hepatic impairment or other conditions that predispose to lactic acidosis.
* History of acute myocardial infarction in the last 6 months
* Serious illness or psychiatric condition.
* Current participation in other protocols with experimental drugs.
* Suspicion of dihidropirimida dehydrogenase(DPD)deficiency.
* Presence of active infection.
* No ability to ingest food orally.
* Patients with metastatic disease to CNS.
* Patients who underwent major surgery in the last 4 weeks.
* Patients who received chemotherapy in the last three weeks.
* Patients who underwent radiotherapy in the last 2 weeks or who received radiotherapy in the target lesion, if this is the only target lesion.
* Patients using oral anticoagulation (warfarin).
* Pregnant or lactating patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate according to RECIST 1.1 | From randomization of the first subject until the database cut-off approximately 12 months later (01Nov2012 up to 01Nov2015). Tumor assessed at 8 week intervals

SECONDARY OUTCOMES:
Progression-free Survival | From randomization of the first subject until the database cut-off approximately 12 months later (01Nov2012 up to 01Nov2015). Tumor assessed at 4 week intervals.
  defined as time from randomization to death from any cause, or even radiological detection/or clinical of disease progression, increased CEA will not be considered isolated progression.
Overall Survival | From randomization of the first subject until the database cut-off approximately 12 months later (01Nov2012 up to 01Nov2015). Tumor assessed at 4 week intervals
  defined as time from first dose of treatment until death, with date of last visit being considered censorship
Adverse Events | From randomization of the first subject until the database cut-off approximately 12 months later (01Nov2012 up to 01Nov2015). Tumor assessed at 4 week intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Do Cancer Do Estado de São Paulo, São Paulo, São Paulo, Brazil